CLINICAL TRIAL: NCT02443623
Title: Vaccinia Vaccination (ACAM2000®) of Plasma Donors for the Production of Vaccinia Immune Globulin Intravenous (VIGIV)
Brief Title: VA-008 ACAM2000® Vaccination of Plasma Donors for the Production of VIGIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VA-008
Record Dates: First submitted 2015-05-06; First posted 2015-05-14 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox Vaccine Adverse Reaction
MeSH Terms: interventions — Vaccination; ACAM2000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Vaccinated with ACAM2000 (Experimental): * To vaccinate plasma donors with the ACAM2000 smallpox vaccine thereby inducing an immune response resulting in high anti-vaccinia antibody titers. The collection of donor plasma will be used in the manufacturing of Vaccinia Immune Globulin Intravenous (VIGIV).
  * To ensure the safety of plasma donors vaccinated with ACAM2000 through the implementation of risk factor screening procedures and the collection of post-vaccination safety data.
  Interventions: Biological: Vaccination with ACAM2000

INTERVENTIONS:
Biological: Vaccination with ACAM2000 — In this study (VA-008), healthy adult male and female volunteers who meet the requirements for source plasma donors and study entry criteria will be vaccinated with the ACAM2000 smallpox vaccine for collection of plasma to be used in the manufacture of VIGIV. There are possible risks associated with ACAM2000 vaccination. To ensure the safety of plasma donors, risk factor screening procedures and the collection of post-vaccination safety data will be assessed throughout the study.

SUMMARY:
Objectives:

* To vaccinate plasma donors with the ACAM2000 smallpox vaccine thereby inducing an immune response resulting in high anti-vaccinia antibody titers. The collection of donor plasma will be used in the manufacturing of Vaccinia Immune Globulin Intravenous (VIGIV).
* To ensure the safety of plasma donors vaccinated with ACAM2000 through the implementation of risk factor screening procedures and the collection of post-vaccination safety data.

DETAILED DESCRIPTION:
This protocol is being conducted to vaccinate plasma donors with the ACAM2000 smallpox vaccine thereby inducing an immune response resulting in high anti-vaccinia antibody titers. The collection of donor plasma will be used in the manufacturing of Vaccinia Immune Globulin Intravenous (VIGIV). The objective of this protocol is to ensure the safety of plasma donors vaccinated with ACAM2000 through the implementation of risk factor screening procedures and the collection of post-vaccination safety data.

Participants will be followed for the duration of the study, an expected average of 90 days as described below in the planned study assessments.

Screening [complete within 14 days before Baseline (Day 0)]:

* Informed consent obtained from prospective donors
* Post-consent information including medical history, smallpox vaccination history, current medications, detailed demographics, BMI, physical exam, vital signs, and assessment for pericarditis/myocarditis symptoms, blood samples will be collected and a baseline EKG (if applicable).

Baseline (Day 0) prior to vaccination:

-Physical exam and vital signs, urine pregnancy test for all female subjects of child-bearing potential, current medications, assessment for pericarditis/myocarditis.

Baseline (Day 0) vaccination and post-vaccination:

-Vaccination with ACAM2000, vaccination site inspection 30 post-vaccination, unanticipated problems, all adverse events including all cardiovascular adverse events (symptoms and signs), concomitant medications.

Post-vaccination Day 3 (±1):

-Assessment for pericarditis/myocarditis, vaccination site inspection, unanticipated problems, unexpected and serious adverse reactions or complications post-vaccination, all adverse events including all cardiovascular adverse events (symptoms and signs).

Post-vaccination Day 7 (±1):

-Assessment of pericarditis/myocarditis symptoms, urine pregnancy test, vaccination site inspection, unanticipated problems, all adverse events including all cardiovascular adverse events (symptoms and signs), concomitant medications.

Post-vaccination Day 12 (±2), 21 (±3), and 28 (±3):

-Assessment of pericarditis/myocarditis symptoms, urine pregnancy test, vaccination site inspection, unanticipated problems, all adverse events including all cardiovascular adverse events (symptoms and signs), concomitant medications.

End of study post-vaccination Day 35 (±3) or Early Withdrawal:

Vital signs, assessment of pericarditis/myocarditis symptoms, urine pregnancy test, vaccination site inspection, unanticipated problems, all adverse events including all cardiovascular adverse events (symptoms and signs), concomitant medications.

Final Safety Assessment Day 90 (±3):

Assessment for pericarditis/myocarditis, unanticipated problems, unexpected and serious adverse reactions or complications post-vaccination, all adverse events including all cardiovascular adverse events (symptoms and signs).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age 18 to 65.
* Normal and healthy (immune competent) as determined by medical history, physical exam, vital signs and clinical laboratory tests during the screening period.
* If all lab results for quantitative IgA immunoglobulin level are lower than 15% below normal range, the subject may not proceed further in the screening process.
* Subject must meet all required subject suitability criteria that pertain to normal source plasma donors.
* Negative HIV serology during screening period.
* Subject must have been previously immunized for smallpox, at ≥3 years prior to commencement of screening assessments, and vaccination history must be confirmed by oral or written history and the presence of a visible pathognomonic smallpox vaccination scar.

Exclusion Criteria:

* History of severe related adverse event(s) from previous participation in VA-001 or VA-006 trials or to any smallpox vaccination.
* The subject, or a household contact or other close/intimate contact of the subject has ANY of the following:

  * Eczema, history of eczema, exfoliative skin conditions, wounds, burns, or other skin conditions at the investigator's discretion.
  * A history of immunodeficiency.
  * Currently or has recently received radiotherapy or chemotherapy, adrenocorticotropic hormone (ACTH), corticosteroids, or immunosuppressive drugs.
  * Eye disease treated with topical steroids.
  * Known or suspected disorders of immunoglobulin synthesis.
  * Leukemia, lymphomas of any type, melanoma, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
  * Has been diagnosed with cancer and who will be undergoing chemotherapy or radiation therapy during the vaccination healing time.
  * Is a transplant recipient (except for corneal transplant).
  * Is pregnant, planning pregnancy or breast feeding (female subjects of childbearing potential must have negative pregnancy test prior to vaccination). Women of child-bearing potential (WOCBP) are temporarily excluded due to COVID.
* Household or other close/intimate contact(s) under the age of 12 months.
* History of allergies to phenol, any of the antibiotics listed in the vaccine content, or any other component of ACAM2000 or its diluents.
* Subjects with kidney disease (except kidney stones).
* Subjects with abnormal EKG at screening (if applicable). To mitigate the risk of enrolling at risk subjects and potentially jeopardizing subject safety an EKG will be performed prior to vaccination with ACAM2000 smallpox vaccine in all potential subjects ≥50 years old and for all potential subjects <50 with two cardiac risk factors as listed immediately below including; severely or morbidly obese or higher obesity classification (BMI ≥36); high blood pressure; high blood cholesterol; diabetes or high blood sugar; a first degree relative who had a heart condition before the age of 50; and current tobacco smokers.
* Subject has three or more of the following risk factors:

  * Severely or morbidly obese or higher obesity classification (BMI ≥36)
  * High blood pressure diagnosed by a doctor
  * High blood cholesterol diagnosed by a doctor
  * Diabetes or high blood sugar diagnosed by a doctor
  * A first degree relative (for example, mother, father, brother, sister) who had a heart condition before the age of 50
  * Currently smokes tobacco (cigarettes)
* Cardiovascular disease or heart condition diagnosed by a doctor at any time in the past, with or without symptoms, including:

  * Arrhythmia
  * Syncope related to cardiac disease
  * Previous myocardial infarction
  * Angina
  * Coronary artery disease
  * Congestive heart failure
  * Cardiomyopathy
  * Stroke or transient ischemic attack
  * Myocarditis
  * Pericarditis
  * Chest pain or shortness of breath with activity (such as climbing stairs), peripheral edema, heart palpitations, dry cough, irregular heartbeat, excessive fatigue, unexplained syncope
  * Other heart conditions being treated by a physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3032 (Actual)
Dates: Start 2015-09; Primary Completion 2021-07 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hall, PhD, Study Director — Emergent BioSolutions
Locations (1):
- Bio Products Laboratory Ltd (plasma vendor of Emergent BioSolutions), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Vaccinated With ACAM2000: Healthy adult male and female volunteers who met the requirements for source plasma donation and study entry criteria were vaccinated with the ACAM2000 smallpox vaccine for collection of plasma to be used in the manufacture of VIGIV. There are possible risks associated with ACAM2000 vaccination. To ensure the safety of plasma donors, risk factor screening procedures and the collection of post-vaccination safety data were assessed throughout the study.
Period: Overall Study
Arm/Group | Single Arm Vaccinated With ACAM2000
Started | 3032
Completed | 2788
Not Completed | 244

BASELINE CHARACTERISTICS:
Population: The safety population consisted of 3032 participants who were vaccinated, including 208 participants who were vaccinated twice (n= 208 includes two participants who were inadvertently vaccinated twice were included twice in demography and all participant counts).
Groups:
- Single Arm Vaccinated With ACAM2000: Healthy adult male and female volunteers who met the requirements for source plasma donation and study entry criteria were vaccinated with the ACAM2000 smallpox vaccine for collection of plasma used in the manufacture of VIGIV.
Arm/Group | Single Arm Vaccinated With ACAM2000
Number analyzed (Participants) | 3032
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 3013
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 765
  Male | 2267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 626
  Not Hispanic or Latino | 2325
  Unknown or Not Reported | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 64
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 13
  Black or African American | 744
  White | 2123
  More than one race | 27
  Unknown or Not Reported | 36
Region of Enrollment [Number; unit: participants]
  United States | 3032
Height [Mean (Standard Deviation); unit: cm] | 174.3 (9.5)
Weight [Mean (Standard Deviation); unit: kg] | 92.5 (20.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccinated Participants With Adverse Events (AEs) Including Serious Adverse Events (SAEs)
Description: Number of subjects with AEs including SAEs up to 90 days after vaccination.
Time Frame: Adverse event data was collected from vaccinated participants through Day 90.
Population: The safety population consisted of 3032 participants who were vaccinated, including 208 participants who were vaccinated twice (n= 208 includes two participants who were inadvertently vaccinated twice and were included twice in demography and all participant counts).
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Vaccinated With ACAM2000
Number analyzed (Participants) | 3032
Participants | 1420

2. Primary Outcome: Number of Vaccinated Participants With Related Adverse Events
Description: Number of subjects with related AEs up to 90 days after vaccination.
Time Frame: Adverse event data was collected from vaccinated participants through Day 90.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Vaccinated With ACAM2000
Number analyzed (Participants) | 3032
Participants | 1190

3. Primary Outcome: Number of Vaccinated Participants With Serious Adverse Events (SAEs)
Description: Number of subjects with SAEs up to 90 days after vaccination.
Time Frame: Adverse event data was collected from vaccinated participants through Day 90.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Vaccinated With ACAM2000
Number analyzed (Participants) | 3032
Participants | 25

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from vaccinated participants through Day 90.
Description: All AEs were elicited by the PI. The causality of an AE was determined by the PI. Diary cards were utilized to help subjects record and track AEs between study assessments. All AEs/reactions on diary cards were reviewed with subjects by the PI and/or designate at the regularly scheduled visits. AEs from the diary card were entered into the data capture (EDC) system. Related AEs are reported under Other (Not Including Serious) AEs;related events were not reported for All-Cause Mortality and SAEs.
Groups:
- Single Arm Vaccinated With ACAM2000 With AEs: Healthy adult male and female volunteers who met the requirements for source plasma donation and study entry criteria were vaccinated with the ACAM2000 smallpox vaccine for collection of plasma used in the manufacture of VIGIV.
- Single Arm Vaccinated With ACAM2000 With Related AEs: Healthy adult male and female volunteers who met the requirements for source plasma donation and study entry criteria were vaccinated with the ACAM2000 smallpox vaccine for collection of plasma used in the manufacture of VIGIV with related adverse events.
Arm/Group | Single Arm Vaccinated With ACAM2000 With AEs | Single Arm Vaccinated With ACAM2000 With Related AEs
All-Cause Mortality (participants affected / at risk) | 1/3032 | 0/0
Serious Adverse Events (participants affected / at risk) | 25/3032 | 0/0
Other Adverse Events (participants affected / at risk) | 1413/3032 | 1190/3032
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Vaccinated With ACAM2000 With AEs (N=3032) | Single Arm Vaccinated With ACAM2000 With Related AEs (N=0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | NA
Acute myocardial infarction (Cardiac disorders) | 1 (1) | NA
Angina pectoris (Cardiac disorders) | 1 (1) | NA
Chest pain (General disorders) | 2 (2) | NA
Non-cardiac chest pain (General disorders) | 2 (2) | NA
Hypersensitivity (Immune system disorders) | 1 (1) | NA
Appendicitis (Infections and infestations) | 1 (1) | NA
Peritonsillar abscess (Infections and infestations) | 1 (1) | NA
Post vaccination autoinoculation (Infections and infestations) | 1 (1) | NA
Upper respiratory tract infection (Infections and infestations) | 1 (1) | NA
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | NA
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | NA
Back injury (Injury, poisoning and procedural complications) | 1 (1) | NA
Head injury (Injury, poisoning and procedural complications) | 1 (1) | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | NA
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Alcoholic seizure (Nervous system disorders) | 1 (1) | NA
Ischaemic stroke (Nervous system disorders) | 1 (1) | NA
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | NA
Syncope (Nervous system disorders) | 1 (1) | NA
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | NA
Bipolar disorder (Psychiatric disorders) | 1 (1) | NA
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Vaccinated With ACAM2000 With AEs (N=3032) | Single Arm Vaccinated With ACAM2000 With Related AEs (N=3032)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 (12) | 8 (9)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear discomort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 1 (1)
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (2) | 0 (0)
Eye pruritus (Eye disorders) | 3 (4) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Scleral hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 24 (24) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (37) | 8 (8)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (18) | 4 (4)
Asthenia (General disorders) | 6 (6) | 4 (4)
Axillary pain (General disorders) | 7 (8) | 5 (5)
Chest discomfort (General disorders) | 10 (11) | 3 (3)
Chest pain (General disorders) | 13 (14) | 0 (0)
Chills (General disorders) | 12 (12) | 6 (6)
Fatigue (General disorders) | 48 (53) | 15 (15)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 15 (17) | 1 (1)
Infusion site hypoaesthesia (General disorders) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0)
Injection site scab (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 23 (23) | 11 (11)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 56 (59) | 32 (34)
Swelling (General disorders) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 1 (1) | 1 (1)
Vaccination site discharge (General disorders) | 1 (1) | 1 (1)
Vaccination site discomfort (General disorders) | 1 (1) | 1 (1)
Vaccinatination site erythema (General disorders) | 2 (2) | 2 (2)
Vaccination site injury (General disorders) | 1 (1) | 1 (1)
Vaccination site irritation (General disorders) | 3 (3) | 3 (3)
Vaccination site joint erythema (General disorders) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 46 (47) | 43 (44)
Vaccination site pruritus (General disorders) | 22 (22) | 21 (21)
Vaccination site rash (General disorders) | 2 (2) | 2 (2)
Vaccination site reaction (General disorders) | 4 (4) | 4 (4)
Vaccination site scab (General disorders) | 1098 (1103) | 1089 (1094)
Vaccination site streaking (General disorders) | 3 (3) | 3 (3)
Vaccination site swelling (General disorders) | 3 (3) | 3 (3)
Vaccination site warmth (General disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 13 (15) | 1 (1)
Smoke sensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 21 (22) | 2 (2)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1)
Post vaccination autoinoculation (Infections and infestations) | 5 (5) | 5 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Vaccination site infection (Infections and infestations) | 2 (2) | 2 (2)
Viral supper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 9 (10) | 9 (10)
Wound (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Blood cholesterol increased (Investigations) | 3 (3) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 0 (0)
Body temperature decreased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (1)
HIV test positive (Investigations) | 2 (2) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 3 (3) | 0 (0)
Heart rate irregular (Investigations) | 3 (4) | 1 (1)
Hepatitis C virus test positive (Investigations) | 1 (1) | 0 (0)
Treponema test positive (Investigations) | 6 (6) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (28) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (12) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 18 (18) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 182 (242) | 58 (63)
Hypoesthesia (Nervous system disorders) | 2 (3) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 6 (7) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Sinus headache (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Affect liability (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0)
Irritability (Psychiatric disorders) | 5 (5) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (50) | 7 (8)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 5 (5)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Application site acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Ovarian cystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0)
Vasectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 5 (5) | 1 (1)
Hypertension (Vascular disorders) | 9 (9) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02443623/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT02443623/SAP_001.pdf